CLINICAL TRIAL: NCT02866669
Title: Collaboration to Improve Blood Pressure in the US Black Belt-addressing the Triple Threat
Brief Title: Southeastern Collaboration to Improve Blood Pressure Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Andrea Cherrington, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: X160722009
Record Dates: First submitted 2016-06-13; First posted 2016-08-15 (Estimated); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Enhanced usual care (Active Comparator): Practices in the usual enhanced care arm will receive a blood pressure medication algorithm developed using national guidelines and content experts on our study team. Practices will be provided the Joint National Committee (JNC) recommended protocol to measuring blood pressures. Practices will receive a laptop workstation that has access to the Patient Activated Learning System - an online education video system.
  Interventions: Behavioral: Enhanced usual care
- Practice facilitation (Experimental): Practices that are randomized to the practice facilitation arm will work with a practice facilitator that will help practice staff for 15 months to make practice level changes to improve hypertension control. Practice facilitation is a highly customized, staged approach to helping a practice to implement process and structural changes to enhance the quality of care and improve patient and staff satisfaction
  Interventions: Behavioral: Practice Facilitation; Behavioral: Enhanced usual care
- Peer coach (Experimental): Participants enrolled from practices that are randomized to the peer coach arm will be matched with peer advisors who will work with the participants for 12 months.
  Interventions: Behavioral: Peer Coach; Behavioral: Enhanced usual care
- Peer coach and Practice facilitation (Experimental): Practices that are randomized to the practice facilitation arm will work with a practice facilitator that will help practice staff for 15 months to make practice level changes to improve hypertension control. The patients will also be matched with peer advisors who will work with the participants for 12 months.
  Interventions: Behavioral: Practice Facilitation; Behavioral: Peer Coach; Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: Practice Facilitation — ractices that are randomized to the practice facilitation arm will work with a practice facilitator that will help practice staff for 15 months to make practice level changes to improve hypertension control. Practice facilitation is a highly customized, staged approach to helping a practice to implement process and structural changes to enhance the quality of care and improve patient and staff satisfaction
  Arms: Peer coach and Practice facilitation; Practice facilitation
Behavioral: Peer Coach — Participants enrolled from practices that are randomized to the peer coach arm will be matched with peer advisors who will work with the participants for 12 months.
  Other Names: Taking Control of Your Health
  Arms: Peer coach; Peer coach and Practice facilitation
Behavioral: Enhanced usual care — Practices in the usual enhanced care arm will receive a blood pressure medication algorithm developed using national guidelines and content experts on our study team. Practices will be provided the Joint National Committee (JNC) recommended protocol to measuring blood pressures. Practices will receive a laptop workstation that has access to the Patient Activated Learning System - an online education video system.

SUMMARY:
The central objective of this proposal is to rigorously compare two strategies designed to improve BP control in primary care practices serving rural Southeastern African Americans with low socioeconomic status (SES) living in the "Black Belt".

In year 1, we're engaging community members (community members who have experience being community peer advisors or have high blood pressure) to develop the study interventions and protocols. In years 2-5, the investigators will test the interventions.

Year 2-5, Aim 3: Enroll 80 practices and 25 African American patients with uncontrolled HTN at each practice (total n=2000) in a cluster-randomized, controlled, 4-arm pragmatic implementation trial to evaluate the three multi- component, multi-level functional interventions finalized in the UH2 phase compared with enhanced usual care.

The study's 4 arms are:

1. Enhanced Usual Care: Practices are provided with educational materials and tools to enhance patient care
2. Peer Coaching: Patients enrolled in these practices will be matched with a peer coach. The peer coach helps the patient to set goals around self-management, including medications, home monitoring, and diet and exercise, and she helps the patient to strategize how to accomplish the goals, using motivational interviewing techniques
3. Practice Facilitation: Practices randomized to this arm will work with a practice facilitator. Practice facilitation is a highly customized, staged approach to helping a practice to implement process and structural changes to enhance the quality of care and improve patient and staff satisfaction
4. Peer coaching and practice facilitation: Practices randomized to this arm will receive both the peer coach intervention and the practice facilitation intervention. Practice facilitators and peer coaches will receive the same training for this hybrid intervention, but the practice facilitator change packet will add examples of activities that integrate peer coaches.

ELIGIBILITY:
Inclusion Criteria:

* African American adults aged 19-85 years
* Uncontrolled HTN, defined as BP >140/90 mm Hg at the time of study enrollment
* Black Belt resident
* English speaking
* Willing to work with a peer coach
* Willing to sign informed consent

Exclusion Criteria:

* Plans to move out of the area within the next two years
* Advanced illness with limited life expectancy
* Pregnant or plans to get pregnant in the next year
* Advanced chronic kidney disease (estimated glomerular filtration rate <45 ml/min/1.73 m2)
* Unwillingness to work with a peer coach or to sign informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1592 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Alabama At Birmingham, Birmingham, Alabama
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Safford MM, Cummings DM, Halladay JR, Shikany JM, Richman J, Oparil S, Hollenberg J, Adams A, Anabtawi M, Andreae L, Baquero E, Bryan J, Sanders-Clark D, Johnson E, Richman E, Soroka O, Tillman J, Cherrington AL. Practice Facilitation and Peer Coaching for Uncontrolled Hypertension Among Black Individuals: A Randomized Clinical Trial. JAMA Intern Med. 2024 May 1;184(5):538-546. doi: 10.1001/jamainternmed.2024.0047. PMID 38497987
- [Derived] Sutton KF, Richman EL, Rees JR, Pugh-Nicholson LL, Craft MM, Peaden SH, Soroka O, Mackey M, Cummings DM, Cherrington AL, Safford MM, Halladay JR; Southeastern Collaboration to Improve Blood Pressure Writing Group. Implementing practice facilitation in research: how facilitators spend their time guiding practices to improve blood pressure control. Implement Sci Commun. 2023 Jul 31;4(1):89. doi: 10.1186/s43058-023-00470-y. PMID 37525267
- [Derived] Shikany JM, Safford MM, Cherrington AL, Halladay JR, Anabtawi M, Richman EL, Adams AD, Holt C, Oparil S, Soroka O, Cummings DM. Recruitment and retention of primary care practices in the Southeastern Collaboration to Improve Blood Pressure Control. Contemp Clin Trials Commun. 2023 Jan 16;32:101059. doi: 10.1016/j.conctc.2023.101059. eCollection 2023 Apr. PMID 36718176
- [Derived] Cummings DM, Adams A, Patil S, Cherrington A, Halladay JR, Oparil S, Soroka O, Ringel JB, Safford MM. Treatment Intensity, Prescribing Patterns, and Blood Pressure Control in Rural Black Patients with Uncontrolled Hypertension. J Racial Ethn Health Disparities. 2023 Oct;10(5):2505-2512. doi: 10.1007/s40615-022-01431-2. Epub 2022 Oct 21. PMID 36271193
- [Derived] Finch AJ, Ringel JB, Dargar S, Halladay J, Cene C, Cherrington A, Cummings D, Safford MM. Greater Social Functioning Associated With Lower Depressive Symptomatology Among Black Belt African Americans Enrolled in the Southeastern Collaboration to Improve Blood Pressure Control Study. Prim Care Companion CNS Disord. 2022 Feb 3;24(1):21m02988. doi: 10.4088/PCC.21m02988. PMID 35114739
- [Derived] Sutton KF, Richman EL, Rees JR, Pugh-Nicholson LL, Craft MM, Peaden SH, Mackey M, Halladay JR; Southeastern Collaboration to Improve Blood Pressure Writing Group. Successful Trial of Practice Facilitation for Plan, Do, Study, Act Quality Improvement. J Am Board Fam Med. 2021 Sep-Oct;34(5):991-1002. doi: 10.3122/jabfm.2021.05.210140. PMID 34535524

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We used a random number generator to randomize practices into 4 trial arms; The goal was to recruit approximately 25 participants at each of the randomized practices. The 4 trial arms were enhanced usual care, practice facilitation, peer coaching, and both practice facilitation and peer coaching. Each participant had baseline, 6 month and 12 month data collected. The intervention duration was one year.
Units Other Than Participants: Practices
Period: Overall Study
Arm/Group | Enhanced Usual Care | Practice Facilitation | Peer Coach | Peer Coach and Practice Facilitation
Started (Practices Randomized) | 406; 18 Practices | 382; 16 Practices | 424; 19 Practices | 380; 16 Practices
Completed | 342; 16 Practices | 260; 12 Practices | 332; 17 Practices | 275; 15 Practices
Not Completed | 64; 2 Practices | 122; 4 Practices | 92; 2 Practices | 105; 1 Practices

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Usual Care | Practice Facilitation | Peer Coach | Peer Coach and Practice Facilitation | Total
Number analyzed (Participants) | 342 | 260 | 332 | 275 | 1209
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (12) | 56 (11) | 58 (12) | 57 (12) | 58 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206 | 153 | 205 | 184 | 748
  Male | 136 | 107 | 127 | 91 | 461
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 7 | 16 | 13 | 51
  Not Hispanic or Latino | 327 | 251 | 316 | 261 | 1155
  Unknown or Not Reported | 0 | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 342 | 260 | 332 | 275 | 1209
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: NC | 182 | 158 | 134 | 145 | 619
  United States: AL | 160 | 102 | 198 | 130 | 590
Baseline systolic BP, mm Hg [Mean (Standard Deviation); unit: mm Hg] | 158 (18) | 156 (17) | 153 (14) | 157 (17) | 156 (16)
Educational Attainment less than high school [Count of Participants; unit: Participants] — Population: One participant was missing information on educational attainment.
  Participants
    number analyzed (Participants) | 342 | 260 | 331 | 275 | 1208
    (all) | 81 | 63 | 64 | 60 | 268
Annual Household Income [Count of Participants; unit: Participants]
  Less than 20K | 141 | 139 | 146 | 121 | 547
  Greater thank 20K | 148 | 84 | 138 | 117 | 487
  Declined/Don't know | 53 | 37 | 48 | 37 | 175
Married [Count of Participants; unit: Participants] — Population: Some participants are missing information on marital status.
  Participants
    number analyzed (Participants) | 340 | 260 | 331 | 273 | 1204
    (all) | 137 | 89 | 110 | 99 | 435
Without Health Insurance [Count of Participants; unit: Participants] | 51 | 56 | 52 | 35 | 194
Has Diabetes [Count of Participants; unit: Participants] | 160 | 123 | 161 | 124 | 568
History of Stroke [Count of Participants; unit: Participants] | 28 | 27 | 32 | 24 | 111
General Self-Reported Health [Count of Participants; unit: Participants]
  Excellent | 6 | 5 | 7 | 3 | 21
  Very Good | 45 | 28 | 41 | 44 | 158
  Good | 141 | 97 | 128 | 98 | 464
  Fair | 128 | 101 | 134 | 106 | 469
  Poor | 22 | 29 | 22 | 24 | 97
Moderate to severe depression (PHQ-8 score >10) [Count of Participants; unit: Participants] — Personal Health Questionnaire Depression Scale (PHQ-8). The scale is comprised of 8 items each of which is scored 0-3. Items are summed up to create a total score ranging from 0-24 with higher scores indicating more worse outcomes and more depressive symptoms. Population: Some participants are missing information on depressive symptoms.
  Participants
    number analyzed (Participants) | 342 | 259 | 331 | 275 | 1207
    (all) | 53 | 59 | 89 | 52 | 253
Someone helps read written materials from the doctor a little to all of the time [Count of Participants; unit: Participants] — Population: Some participants were missing information on health literacy.
  Participants
    number analyzed (Participants) | 342 | 259 | 331 | 273 | 1205
    (all) | 132 | 120 | 109 | 94 | 455
Problems learning about conditions because can't understand written info. [Count of Participants; unit: Participants] — Has problems learning about conditions because can't understand written info a little to all of the time. Population: Some participants were missing information on health literacy
  Participants
    number analyzed (Participants) | 341 | 258 | 329 | 274 | 1202
    (all) | 123 | 132 | 121 | 99 | 475
Reported greater than 1 barrier to medication adherence [Count of Participants; unit: Participants] — Population: Some participants are missing information on barriers to medication adherence.
  Participants
    number analyzed (Participants) | 334 | 259 | 322 | 269 | 1184
    (all) | 262 | 212 | 262 | 225 | 961
Social Isolation score (PROMIS) [Median (Inter-Quartile Range); unit: score on a scale] — We measured isolation using the Patient Reported Outcomes Measurement Information System (PROMIS) short-form social functioning scale. To each question subjects were asked to respond with "never," "rarely," "sometimes," "usually," or "always." A numerical value was attached to each of these answers, ranging from 1 ("never") to 5 ("always"). Raw scores were translated to standardized t-scores to allow comparison of our sample to the U.S population. The scale is comprised of 4 items. Raw scores range from 0-20 and scale scores range from 34.8-74.2. Higher scores indicate greater isolation. Population: Some participants are missing information on social isolation
  score on a scale
    number analyzed (Participants) | 340 | 254 | 328 | 274 | 1196
    (all) | 43 [35 to 52] | 48 [35 to 56] | 48 [35 to 54] | 43 [35 to 52] | 46 [35 to 54]
Baseline perceived emotional support score (PROMIS) [Median (Inter-Quartile Range); unit: score on a scale] — We measured perceived emotional support using the Patient Reported Outcomes Measurement Information System (PROMIS) short-form social functioning scale. For 4 questions, participants were asked to respond with "never," "rarely," "sometimes," "usually," or "always." A numerical value was attached to each of these answers, ranging from 1 ("never") to 5 ("always"). Raw scores were translated to standardized t-scores to allow comparison of our sample to the U.S population. Raw scores ranged from 4-20 and scale scores ranged from 25.7-62 with higher scores indicating greater emotional support. Population: Participants were missing information on perceived emotional support
  score on a scale
    number analyzed (Participants) | 341 | 259 | 331 | 275 | 1206
    (all) | 62 [49 to 62] | 53 [44 to 62] | 53 [44 to 62] | 62 [47 to 62] | 56 [45 to 62]
Perceived Instrumental Support score (PROMIS) [Median (Inter-Quartile Range); unit: score on a scale] — We measured perceived instrumental support using the Patient Reported Outcomes Measurement Information System (PROMIS) short-form social functioning scale. For 4 questions, subjects were asked to respond with "never," "rarely," "sometimes," "usually," or "always." A numerical value was attached to each of these answers, ranging from 1 ("never") to 5 ("always"). Raw scores were translated to standardized t-scores to allow comparison of our sample to the U.S population. Raw scores ranged from 4-20. Scale scores ranged from 29.3-69.3 with a higher score indicating greater instrumental support. Population: Some participants were missing information on perceived instrumental support
  score on a scale
    number analyzed (Participants) | 337 | 256 | 325 | 270 | 1188
    (all) | 63 [51 to 63] | 54 [47 to 63] | 63 [49 to 63] | 63 [51 to 63] | 63 [49 to 63]
Perceived Stress Scale [Median (Inter-Quartile Range); unit: score on a scale] — The 4-item Cohen's perceived stress scale that is measured on a 5-point scale (0 = never, 1= almost never, 2 = sometimes, 3 = fairly often and 4- very often). Items 2 and 3 are reverse coded and then all for items are summed to created a total score that ranges from 0 -16. A higher score is negative indicating greater perceived stress. Population: Some participants were missing information on stress
  score on a scale
    number analyzed (Participants) | 336 | 256 | 330 | 274 | 1196
    (all) | 4 [1 to 7] | 6 [2 to 8] | 6 [2 to 8] | 5 [2 to 8] | 5 [2 to 8]
Patient Assessment of Chronic Illness Care (PACIC) [Mean (Standard Deviation); unit: score on a scale] — Patient Assessment of Care for Chronic Conditions (PACIC) measures how patients perceive their chronic condition(s) are being managed by their health care team. Patients fill out a survey of 20 questions regarding the care of their chronic condition(s) over the last 12 months. Responses use a Likert scale from 1-5, where 1 signifies "None of the time" and 5 signifying "Always". PACIC was scored by summing participants' responses across all 20 items then dividing by 20. The range of total score is 1-5 with higher scores indicating better perceived chronic condition care. Population: Some participants are missing information on the PACIC
  score on a scale
    number analyzed (Participants) | 318 | 243 | 317 | 261 | 1139
    (all) | 3 (1) | 3 (1) | 3 (1) | 3 (1) | 3 (1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Blood Pressure Control (Systolic Pressure Less Than 140 mm Hg and Diastolic Pressure Less Than 90 mm Hg) at 12 Months
Description: Blood pressure (BP) control is defined as systolic pressure less than 140 mm Hg and diastolic pressure less than 90 mm Hg. Difference in BP control at 12 month follow-up between trial arms. BP was assessed in the practice by a research assistant using a standardized protocol at baseline, 6, and 12 months.
Time Frame: 12 months
Population: There are 4 arms in this study. Arm one is enhanced usual care. Arm 2 is practice facilitation. Arm 3 is peer coaching. In arm 4 practices received practice facilitation and participants peer coaching. Numbers will be different from final numbers in flow diagram because final sample includes participants that had 6 month or 12 month BP data.
Measure: Number; unit: participants
Arm/Group | Enhanced Usual Care | Practice Facilitation | Peer Coach | Peer Coach and Practice Facilitation
Number analyzed (Participants) | 309 | 241 | 309 | 254
participants | 112 | 87 | 130 | 92

2. Secondary Outcome: Change in Systolic Blood Pressure Between Baseline and 12 Months
Description: Change in systolic blood pressure between baseline and 12 months, which is analyzed by subtracting the baseline systolic BP from the 12 month systolic BP.
Time Frame: 12 months
Population: There are 4 arms in this study. Arm one is enhanced usual care. Arm 2 is practice facilitation. Arm 3 is peer coaching. In arm 4 practices received practice facilitation and participants peer coaching.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Enhanced Usual Care | Practice Facilitation | Peer Coach | Peer Coach and Practice Facilitation
Number analyzed (Participants) | 309 | 241 | 309 | 254
mm Hg | -11 (23) | -10 (24) | -11 (21) | -12 (22)

3. Secondary Outcome: Change in Satisfaction With Chronic Illness Care Between Baseline and 12 Months
Description: Patient Assessment of Care for Chronic Conditions (PACIC) measures how patients perceive their chronic condition(s) are being managed by their health care team. Patients fill out a survey of 20 questions regarding the care of their chronic condition(s) over the last 12 months. Used a Likert scale from 1-5, where 1 signifies "None of the time" and 5 signifying "Always". PACIC was scored by summing participants' responses across all 20 items then dividing by 20. This score was calculated at baseline and 12 months follow-up. A change in score for each participant was created by subtracting the 12 months follow-up PACIC score from the baseline PACIC score.
Time Frame: 12 months
Population: There are 4 arms in this study. Arm one is enhanced usual care. Arm 2 is practice facilitation. Arm 3 is peer coaching. In arm 4 practices received practice facilitation and participants received peer coaching.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | Practice Facilitation | Peer Coach | Peer Coach and Practice Facilitation
Number analyzed (Participants) | 282 | 223 | 301 | 231
score on a scale | 0 (1) | 0 (1) | 0 (1) | 0 (1)

4. Secondary Outcome: Change in Physical Component Summary Score (PCS) of the Short Form 12 (SF12)
Description: Change in health related quality of life measured using self report scale Short form-12. Six questions comprise the PCS. Of the six questions, one question ranges on a 5 point Likert scale from excellent to poor. Two questions range on a 3 point Likert scale from a lot to not at all. Two questions are dichotomous as yes or no. One question ranges on a 5 point Likert scale from extremely to not at all. Different weights are applied to each item to results in scores ranging from 0-100 with higher scores indicating higher functioning.
Time Frame: 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | Practice Facilitation | Peer Coach | Peer Coach and Practice Facilitation
Number analyzed (Participants) | 314 | 238 | 312 | 251
score on a scale | 2 (9) | 1 (9) | 2 (9) | 2 (10)

5. Secondary Outcome: Change in the Mental Component Summary Score (MCS) From the Short Form 12 (SF12)
Description: Change in health related quality of life measured using self report scale Short form-12. Six questions comprise the MCS. Of the six questions, two questions are dichotomous as yes or no. One question ranges on a 5 point Likert scale from all of the time to none of the time. Three questions range on a 6 point Likert scale from all of the time to none of the time. Different weights are applied to each item to result in a score ranging from 0-100 with higher scores indicating higher mental functioning.
Time Frame: 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | Practice Facilitation | Peer Coach | Peer Coach and Practice Facilitation
Number analyzed (Participants) | 314 | 238 | 312 | 251
score on a scale | 3 (11) | 2 (11) | 3 (12) | 3 (12)

6. Secondary Outcome: Self-reported ED Visit or Evidence of an ED Visit at Chart Review Between Baseline and 6 Months
Description: Outcome was defined by self-reported question (yes/no) or chart review. Those who reported yes to the question, "In the past 6 months have you been seen in an ER/ED but not admitted overnight" were considered having the outcome. Data collectors looked for ED visits in patient's charts between baseline and 6 month visit. The outcome measure timeframe is between baseline and 6 months.
Time Frame: between baseline and 6 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Enhanced Usual Care | Practice Facilitation | Peer Coach | Peer Coach and Practice Facilitation
Number analyzed (Participants) | 334 | 252 | 319 | 269
participants | 90 | 53 | 77 | 65

7. Secondary Outcome: Self-reported ED Visit or Evidence of an ED Visit in Chart Review Between 6 Months and 12 Months
Description: Outcome was defined by self-reported question (yes/no) or chart review. Those who reported yes to the question, "In the past 6 months have you been seen in an ER/ED but not admitted overnight" were considered having the outcome. Data collectors looked for ED visits in patient's charts between their 6 month and 12 month follow-up. The outcome measure timeframe is between 6 months and 12 month follow-up.
Time Frame: between 6 months to 12 month
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Enhanced Usual Care | Practice Facilitation | Peer Coach | Peer Coach and Practice Facilitation
Number analyzed (Participants) | 322 | 246 | 321 | 262
participants | 78 | 59 | 66 | 55

8. Secondary Outcome: Self-reported Hospitalization or Evidence of Hospitalization in Chart Review Between Baseline and 6 Months
Description: Outcome was defined by self-reported question (yes/no) or chart review. Those who reported yes to the question, "In the past 6 months have you been hospitalized overnight?" were considered having the outcome.
  Data collectors looked for hospitalization in patient's charts between baseline and 6 month visit. The outcome measure timeframe is between baseline and 6 months.
Time Frame: between baseline to 6 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Enhanced Usual Care | Practice Facilitation | Peer Coach | Peer Coach and Practice Facilitation
Number analyzed (Participants) | 334 | 252 | 319 | 269
participants | 32 | 29 | 32 | 28

9. Secondary Outcome: Self-Reported Hospitalization or Evidence of Hospitalization in Chart Review Between 6 Month and 12 Month
Description: Outcome was defined by self-reported question (yes/no) or chart review. Those who reported yes to the question, "In the past 6 months have you been hospitalized overnight?" were considered having the outcome. Data collectors looked for hospitalizations in patient's charts between their 6 month and 12 month follow-up. The outcome measure timeframe is between 6 months and 12 month follow-up.
Time Frame: between 6 month to 12 month
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Enhanced Usual Care | Practice Facilitation | Peer Coach | Peer Coach and Practice Facilitation
Number analyzed (Participants) | 322 | 246 | 321 | 262
participants | 24 | 35 | 32 | 30

10. Secondary Outcome: Change in Perceived Stress
Description: The 4-item Cohen perceived stress scale that are measured on a 5-point scale (0 = never, 1= almost never, 2 = sometimes, 3 = fairly often and 4- very often). Items 2 and 3 are reverse coded and then all for items are summed to created a total score that ranges from 0 -16. A higher score is negative indicating greater perceived stress.
Time Frame: 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | Practice Facilitation | Peer Coach | Peer Coach and Practice Facilitation
Number analyzed (Participants) | 314 | 240 | 316 | 251
score on a scale | 0 (3) | -1 (4) | -1 (4) | -1 (4)

11. Other Pre Specified Outcome: Self-reported Stroke
Description: Self-reported stroke was defined as participants reporting yes to the question: Since the last time we spoke, were you ever told by a physician that you had a stroke?
Time Frame: 12 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Enhanced Usual Care | Practice Facilitation | Peer Coach | Peer Coach and Practice Facilitation
Number analyzed (Participants) | 320 | 243 | 319 | 254
participants | 6 | 14 | 5 | 4

12. Other Pre Specified Outcome: Change in Instrumental Support
Description: We measured change in perceived instrumental support between baseline and 12 months using the Patient Reported Outcomes Measurement Information System (PROMIS) short-form social functioning scale. To each question subjects were asked to respond with "never," "rarely," "sometimes," "usually," or "always." A numerical value was attached to each of these answers, ranging from 1 ("never") to 5 ("always"). Raw scores were translated to standardized t-scores to allow comparison of our sample to the U.S population. "). The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Raw scores ranged from 4-20. Scale scores ranged from 29.3-69.3 with a higher score indicating greater instrumental support.
Time Frame: 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Enhanced Usual Care | Practice Facilitation | Peer Coach | Peer Coach and Practice Facilitation
Number analyzed (Participants) | 313 | 242 | 311 | 250
T score | 0 (8) | 2 (9) | 1 (10) | 1 (8)

13. Other Pre Specified Outcome: Change in Perceived Emotional Support
Description: We measured change perceived emotional support between baseline and 12 months using the Patient Reported Outcomes Measurement Information System (PROMIS) short-form social functioning scale. To each question subjects were asked to respond with "never," "rarely," "sometimes," "usually," or "always." A numerical value was attached to each of these answers, ranging from 1 ("never") to 5 ("always"). The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Raw scores were translated to standardized t-scores to allow comparison of our sample to the U.S population. Raw scores ranged from 4-20 and scale scores ranged from 25.7-62 with higher scores indicating greater emotional support.
Time Frame: 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Enhanced Usual Care | Practice Facilitation | Peer Coach | Peer Coach and Practice Facilitation
Number analyzed (Participants) | 317 | 244 | 316 | 253
T score | 0 (8) | 2 (9) | 2 (9) | 2 (10)

14. Other Pre Specified Outcome: Change in Social Isolation
Description: We measured change in isolation between baseline and 12 months using the Social Isolation Patient Reported Outcomes Measurement Information System (PROMIS) short-form social functioning scale. To each question subjects were asked to respond with "never," "rarely," "sometimes," "usually," or "always." A numerical value was attached to each of these answers, ranging from 1 ("never") to 5 ("always"). Raw scores were translated to standardized t-scores to allow comparison of our sample to the U.S population. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. The scale is comprised of 4 items. Raw scores range from 0-20 and scale scores range from 34.8-74.2. Higher scores indicate greater isolation.
Time Frame: 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Enhanced Usual Care | Practice Facilitation | Peer Coach | Peer Coach and Practice Facilitation
Number analyzed (Participants) | 316 | 236 | 311 | 250
T score | -1 (9) | -2 (10) | -2 (10) | -1 (10)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Sample for serious and non-serious adverse events includes only enrolled participants with follow-up data (6 or 12 month data) on blood pressure, chart review, self-reported sides effects and self-reported hospitalizations/ED visits.
  Sample for all-cause mortality includes only enrolled participants with follow-up data (6 or 12 month data) on blood pressure, chart review, self-reported sides effects and self-reported hospitalizations/ED visits OR have an adverse events form.
Arm/Group | Enhanced Usual Care | Practice Facilitation | Peer Coach | Peer Coach and Practice Facilitation
All-Cause Mortality (participants affected / at risk) | 2/344 | 0/284 | 5/335 | 7/284
Serious Adverse Events (participants affected / at risk) | 177/342 | 152/283 | 162/330 | 148/285
Other Adverse Events (participants affected / at risk) | 66/342 | 62/283 | 63/330 | 41/285
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Usual Care (N=342) | Practice Facilitation (N=283) | Peer Coach (N=330) | Peer Coach and Practice Facilitation (N=285)
Any ED Visit (General disorders) | 108 (155) | 81 (120) | 105 (155) | 85 (132)
Any hospitalization (General disorders) | 45 (63) | 44 (57) | 52 (64) | 41 (50)
Self reported falls with Ed visit (General disorders) | 7 (8) | 15 (16) | 8 (8) | 5 (7)
Self reported stroke (General disorders) | 14 (16) | 24 (28) | 8 (10) | 12 (14)
Hypertension (Cardiac disorders) | 55 (66) | 54 (66) | 37 (41) | 44 (49) — Systolic Blood Pressure great than or equal to 180 or diastolic blood pressure great than or equal to 110 (from visit)
Hypotension (Cardiac disorders) | 19 (20) | 9 (10) | 19 (20) | 18 (18) — Systolic blood pressure less than 90 or diastolic blood pressure less than 90 (from visit)
OTHER ADVERSE EVENTS (reported when occurring in more than 05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Usual Care (N=342) | Practice Facilitation (N=283) | Peer Coach (N=330) | Peer Coach and Practice Facilitation (N=285)
Self reported dizziness upon standing or fainting (General disorders) | 22 (23) | 29 (34) | 31 (33) | 26 (27)
Self reported falls that did not result in an ED visit (General disorders) | 47 (56) | 43 (52) | 40 (53) | 20 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT02866669/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT02866669/SAP_001.pdf